CLINICAL TRIAL: NCT05590975
Title: Evaluation of Play & Care Together (PACT) Implementation for Improved Resilience, Life Skills, and Psychosocial Skills Among Participating Children and Peer Supporters
Brief Title: Evaluation of Play and Care Together (PACT) Implementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Right to Play (Other)
Responsible Party: Principal Investigator, Dr Rozina Karmaliani, Professor & Dean, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-7690-22673
Record Dates: First submitted 2022-10-04; First posted 2022-10-21 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Resilience; Psychosocial Wellbeing; Peer Problem
Keywords: Resilience among children; Life skills; Peer social behavior

STUDY DESIGN:
Intervention Model Description: The assessment will be carried out parallel in the intervention and the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer Supporter and Adult coach intervention (Experimental): Intervention group will receive PACT module through peer supporters and adult coaches
  Interventions: Behavioral: PACT Intervention
- Adult coach intervention (Experimental): Intervention group will receive PACT module through adult coaches only
  Interventions: Behavioral: PACT Intervention
- Control Group (No Intervention): Control group will receive PACT intervention after the completion of intervention and evaluation with 1st PACT intervention arm.

INTERVENTIONS:
Behavioral: PACT Intervention — PACT Intervention is a group based session delivered by Peer supporters and adult coaches on PACT module. There will be 10 sessions, one per week for 90 to 120 minutes each.
  Arms: Adult coach intervention; Peer Supporter and Adult coach intervention

SUMMARY:
This study aims to evaluate the effectiveness of PACT intervention in improving resilience, life skills, and psychosocial skills among children and peer supporters. The evaluation will be carried out in the Public Schools of Karachi, Sindh, Pakistan.

DETAILED DESCRIPTION:
Right to Play is a non-governmental organization that offers play-based life skills education in public schools of Pakistan. This project aim to improve psychosocial wellbeing, resilience and social and emotional life skills of students enrolled in secondary schools of Lyari in Karachi South, Sindh, Pakistan through "Play and Act Together (PACT)" curriculum. The Aga Khan University will evaluate effectiveness of their intervention that will be offered in public schools of Karachi. Data will be collected from grade 6 students(children) and grade 7 or 8 peer supporters at baseline, midline and endline of the study. Moreover, throughout PACT intervention, fidelity monitoring would be ensured randomly for 3 sessions out of 10 through a checklist to evaluate accuracy of PACT intervention delivered. Furthermore, feasibility checklist would be filled by each participant at the end of the study to analyze the satisfaction, feasibility of PACT intervention and important learnings from PACT curriculum. After the intervention, focus group discussion will took place to learn about the experiences of children, peer supporters and adult coaches who received PACT intervention.

ELIGIBILITY:
Inclusion Criteria:

* Have not participated in previous Right to Play activities
* Voluntarily agree to participate in this program in 2022-23
* More than 30 students in grades 6 enrolled
* A safe playing area (either indoors or outdoors)
* Only Boy or Only girl school
* Sindh Literacy and Education Department direct administration
* Children of grade 6 age 12-15 years
* Children who give assent to participate
* Parents who give consent to participate their children

Exclusion Criteria:

* Schools who does not give consent to participate
* Children who do not give assent
* Parents who do not give consent

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Grade 6 children Grade 7 and 8 Peer supporters
Enrollment: 212 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Resilience | Baseline ( at the time of enrolment), midline (after 5 weeks) and Endline (within two weeks of intervention)
  Tool: Child and Youth Resilience Measure 28: It is a 28 items scale. Point values are assigned to responses; Not at all=1; A little= 2; Somewhat= 3; Quite a bit= 4; A lot= 5. Sum of all items= Higher scores indicate higher levels of characteristics associated with resilience.
  Cutoff: Scores below 65 indicate low resilience; between 65 and 81 show moderate resilience; above 81 will be interpreted as high levels of resilience 3 subscales: Individual, relationships with primary care-givers, and contextual factors that facilitate a sense of belonging
Change in Resilience | Baseline ( at the time of enrolment), midline (after 5 weeks) and Endline (within two weeks of intervention)
  Tool: Resilience Scale 14: This is a 14-item scale in which point values are assigned to responses: strongly disagree=1-4; strongly agree= 5-7.
  Validated scale in Pakistan Higher scores indicate higher levels of characteristics associated with resilience.
  Its individual resilience scale.
Change in social and emotional life skills | Baseline ( at the time of enrolment), midline (after 5 weeks) and Endline (within two weeks of intervention)
  Multidimensional Scale of Life Skills in Late Childhood: This is a 19 items scale use to assess the different life skills among children. Point values are assigned to responses; Never=1; Rarely= 2; Sometimes= 3; Very often= 4; Always= 5.
  Lower score indicate no skills while higher score indicate good skills.
Change in Peer social behaviour | Baseline ( at the time of enrolment), midline (after 5 weeks) and Endline (within two weeks of intervention)
  Tool: Strengths and Difficulties Questionnaire: Sub scales (Peer Problem Scale, Prosocial Scale) Score: 0-10 for each subscale Cutoff: Minimum score is positive change while maximum score is negative change.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan